CLINICAL TRIAL: NCT02264704
Title: Exercise Intensity and Immune Function in Multiple Sclerosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of the West of Scotland (Other)
Collaborators: National Heatlh Service Ayrshire and Arran (Other Government)
Responsible Party: Principal Investigator, Ryan Bell, Postgraduate Student, University of the West of Scotland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 157624 (Registry Identifier: Integrated Research Application Service (IRAS))
Record Dates: First submitted 2014-10-08; First posted 2014-10-15 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2014-10

CONDITIONS: Multiple Sclerosis
Keywords: MS; Exercise; Training; Multiple sclerosis; Immune response; Neurotrophin; Cytokine; Fatigue
MeSH Terms: conditions — Multiple Sclerosis; Motor Activity; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- High intensity exercise (Experimental): High intensity exercise Participants will exercise at high intensity (70% VO2 peak) intermittently (30 seconds on, 30 seconds off) for 15 minutes, twice weekly for 15 weeks.
  Interventions: Other: High intensity exericse
- Moderate intensity exercise (Experimental): Participants exercise at moderate intensity (35% VO2 peak) continuously for 15 minutes, twice weekly for 15 weeks.
  Interventions: Other: Moderate intensity exericse
- Usual Care (No Intervention): Participants receive usual medical care.

INTERVENTIONS:
Other: High intensity exericse — Participants will exercise at high intensity (70% VO2 peak) intermittently (30 seconds on, 30 seconds off) for 15 minutes, twice weekly for 15 weeks. Workload may increase as the study progresses based on heart rate response.
  Arms: High intensity exercise
Other: Moderate intensity exericse — Participants exercise at moderate intensity (35% VO2 peak) continuously for 15 minutes, twice weekly for 15 weeks. Workload may increase as the study progresses based on heart rate response.
  Arms: Moderate intensity exercise

SUMMARY:
This study aims to determine the effect of exercise intensity within a 15 week programme in moderately disabled people with multiple sclerosis (MS). Although earlier research has shown that exercise is safe and may improve health related factors such as mobility and fatigue, the intensity at which exercise offers the most benefit has not yet been defined.

Participants will be randomly assigned to one of three groups - high intensity, moderate intensity or usual care. Participants in the exercising groups (high and moderate intensity) will take part in a supervised 15 week cycling exercise programme based in the Douglas Grant Rehabilitation Centre. Those assigned to the usual care (control) group will continue to receive their usual medical care and will not participate in the exercise programme. The acute immune response to exercise will also be measured.

Participants from all three groups will be monitored regularly. Clinical outcomes of the study include immunological markers, exercise capacity, mobility, fatigue, quality of life and cognitive ability. These will be measured by a combination of blood tests, physical assessments and questionnaires.

It is hypothesised that high intensity exercise will cause a favourable, anti-inflammatory response which will be associated with greater improvements in physical and psychological outcomes than both moderate intensity exercise and usual care.

DETAILED DESCRIPTION:
Recruited patients will initially undergo baseline measurements including BMI. Neurotrophin (BDNF and NGF) and cytokine (IFN-Y and IL-4) concentration will be measured from participant serum using commercially available ELISA kits (R&D systems).

Assessments of cognitive ability, mood, fatigue and quality of life will also be performed using psychometric tests as described in outcomes. Exercise capacity and mobility will be also be measured.

Participants will also undergo a maximal exercise test, recently validated for use in this patient population (Heine et al., 2014). Briefly, rested participants will initially cycle at a power of 25W whilst maintaining a minimum cadence of 60rpm as a 5 minute warm-up. This leads directly into the testing period, during which the power is increased incrementally (15W per minute) until the point of volitional termination or a drop in cadence of 10rpm below the minimum (60 rpm). Peak oxygen consumption (VO2 peak) is used as a measure of cardiorespiratory fitness.

Participants will be randomly assigned to one of three groups - high intensity (HI), moderate intensity (MI) or usual care (UC). Exercising groups will take part in a 15 week programme. All exercise will be performed on a cycle ergometer and will be carried out twice per week for 15 weeks (30 sessions) at the Douglas Grant Rehabilitation Centre, Irvine. In all sessions HI participants will exercise intermittently (30 seconds on 30 seconds off) at 80% of the peak power (based on maximal exercise test) for 15 minutes. MI participants will exercise continuously at 40% peak power for 15 minutes. To ensure exercise intensity remains consistent throughout the programme the workload will progressively increase over time to accommodate any increases in participant fitness levels as measured by %HR. UC participants will not participate in the supervised exercise programme but will continue to receive their usual care.

5 weeks after completion of the exercise programme, a follow-up testing session will occur.

ELIGIBILITY:
Inclusion Criteria:

* Clinically confirmed MS (according to the revised 2010 McDonald criteria) (Polman et al., 2011)
* Expanded disability status scale (EDSS) 3.0-5.0

Exclusion Criteria:

* Unable to consent due cognitive impairment or mental illness
* Immunomodulatory therapy in past 3 months
* Steroid therapy in the past 6 weeks
* Existence of medical contraindications for exercise i.e. cardiovascular or orthopaedic disease.
* Compounding neurological condition other than MS

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 63 (Estimated)
Dates: Start 2014-11; Primary Completion 2015-07 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Change in serum brain-derived neurotrophic factor (BDNF) level | Chronic - Baseline, week 7, week 15 and follow-up (week 20). Acute - 15 mins, 30 mins and 1 hour post-exercise
  The level of brain-derived neurotrophic factor in participant serum will be determined by analysing blood samples using commercially available ELISA assays.

SECONDARY OUTCOMES:
Change in serum nerve growth factor (NGF) level | Chronic - Baseline, week 7, week 15 and follow-up (week 20). Acute - 15 mins, 30 mins and 1 hour post-exercise
  The level of nerve growth factor in participant serum will be determined by analysing blood samples using commercially available ELISA assays.
Change in serum interleukin-4 (IL-4) level | Chronic - Baseline (week 0), week 7, week 15 and follow-up (week 20). Acute - 15 mins, 30 mins and 1 hour post-exercise
  The level of interleukin-4 in participant serum will be determined by analysing blood samples using commercially available ELISA assays.
Change in serum interferon gamma (IFN-γ) level | Chronic - Baseline (week 0), week 7, week 15 and follow-up (week 20). Acute - 15 mins, 30 mins and 1 hour post-exercise
  The level of interferon gamma in participant serum will be determined by analysing blood samples using commercially available ELISA assays.
Change in mobility | Baseline, weeks 5, 10, 15 and follow up (week 20)
  Participant mobility and balance will be assessed by the timed up and go test (TUG). Individuals safely rise from a standard armchair, walk a distance of 3 metres, turn around and return to a seated position. Usual walking aids may be used however personal assistance is not permitted.
Change in exercise capacity | Baseline, weeks 5, 10, 15 and follow up (week 20)
  Exercise capacity will be assessed by the six minute walk test (6MWT). Participants walk continuously, turning at a defined distance, until six minutes have passed. Total distance travelled is the measured outcome.
Change in fatigue | Baseline, weeks 5, 10, 15 and follow up (week 20)
  Self-reported fatigue will be assessed by the 21 item modified fatigue impact scale (MFIS) which has been previously validated for use in this patient population.
Change in health-related quality of life | Baseline, weeks 5, 10, 15 and follow up (week 20)
  Health-related quality of life will be assessed by the 29 item multiple sclerosis impact scale questionnaire (MSIS-29). MSIS-29 analyses both mental and physical aspects of quality of life.
Change in cognitive ability | Baseline, weeks 5, 10, 15 and follow up (week 20)
  The brief international cognitive assessment for multiple sclerosis (BICAMS) is a short test battery which assesses information processing speed, visual memory and verbal learning ability.
Number of sessions attended | 15 weeks
  Adherence will be measured by number of exercise sessions attended across the 15 week intervention (30 sessions).
Change in cardiorespiratory fitness | Baseline and week 15
  Peak oxygen consumption (VO2 peak) will be measured via a maximal exercise test tailored for this patient population (Heine et al., 2014).
Change in mood | Baseline, weeks 5, 10, 15 and follow up (week 20)
  Mood will be assessed by the hospital anxiety and depression scale (HADS). HADS is a 14 item questionnaire designed to analyse self-reported indicators of anxiety and depression.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Bell, MSc, Principal Investigator — University of the West of Scotland
Locations (1):
- Douglas Grant Rehabilitation Centre, Ayrshire Central Hospital, Irvine, Ayrshire, United Kingdom

REFERENCES:
- [Background] Heine M, Hoogervorst EL, Hacking HG, Verschuren O, Kwakkel G. Validity of maximal exercise testing in people with multiple sclerosis and low to moderate levels of disability. Phys Ther. 2014 Aug;94(8):1168-75. doi: 10.2522/ptj.20130418. Epub 2014 Mar 27. PMID 24677255
- [Background] Collett J, Dawes H, Meaney A, Sackley C, Barker K, Wade D, Izardi H, Bateman J, Duda J, Buckingham E. Exercise for multiple sclerosis: a single-blind randomized trial comparing three exercise intensities. Mult Scler. 2011 May;17(5):594-603. doi: 10.1177/1352458510391836. Epub 2011 Jan 19. PMID 21247971